CLINICAL TRIAL: NCT00975949
Title: Neurodevelopmental Outcomes and Quality of Life and Fluconazole Prophylaxis
Brief Title: Neurodevelopmental Outcomes and Fluconazole Prophylaxis
Acronym: NDFP
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, David A Kaufman, Prinicipal Investigator, University of Virginia
Other Study IDs: 13697
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Neurodevelopmental Outcomes
Keywords: fluconazole prophylaxis; fungal colonization; fungal infection; preterm infants; long term outcomes; quality of life
MeSH Terms: conditions — Mycoses | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fluconazole Group: These subjects received fluconazole in our NICU fluconazole prophylaxis study during 1998-2000
  Interventions: Other: Survey
- Placebo Group: These subjects received a placebo during our NICU fluconazole prophylaxis study during 1998-2000
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Parents of subjects were interviewed and two surveys were obtained, the Child Health Questionnaire and the Vineland-II.

SUMMARY:
The purpose of this study is to compare the neurodevelopmental outcome and quality of life between the fluconazole-treated and the placebo-treated patients that were enrolled in a fluconazole prophylaxis study that occurred in the investigators' neonatal intensive care unit (NICU) between 1998-2000.

DETAILED DESCRIPTION:
Invasive fungal infections in preterm infants is associated with significant morbidity and mortality. Mortality in infected infants < 1000 grams is between 26-66% and neurodevelopmental impairment occurs in 57%.1-13 Between 1998-2000 we conducted a randomized placebo controlled trial of fluconazole prophylaxis in 100 infants <1000 grams at birth(IRB-HSR #9389). Invasive fungal infections occurred in none of the fluconazole-treated patients compared to 20% of the placebo group. Following this study the efficacy has been confirmed in a multicenter randomized controlled trial and 7 retrospective studies. One major issue that has remained is whether the fluconazole-treated infants have better neurodevelopmental outcomes as well as if it is safe without an increase in neurodevelopmental impairment.

Neurodevelopmental outcomes can be assessed by testing and examinations or by parental and child questionnaires. In addition, quality of life is an important context of outcomes. Recent conceptualizations of quality of life recognize the multidimensional nature of quality of life, including psychological and social functioning, consistent with the World Health Organization's definition of health as "not only the absence of disease and infirmity, but the presence of physical, mental, and social well-being." The World Health Organization subsequently emphasized the growing consensus that quality of life is a subjective experience, defined as "individuals' perceptions of their position in life in the context of the culture and value systems in which they live, and in relation to their goals, expectations, standards, and concerns."

To address these issues, we aim to study and compare the neurodevelopmental outcome and quality of life between our fluconazole-treated and placebo-treated patients in our initial study

ELIGIBILITY:
Inclusion Criteria:

* Parents or guardians and their infants who survived and were enrolled in our initial study of fluconazole prophylaxis for prevention of fungal colonization and infection in preterm infants < 1000 grams

Exclusion Criteria:

* Persons not meeting the inclusion criteria

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects were born <1000 grams, treated in our NICU, and are now 7 to 10 years of age.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental impairment and poor quality of life | 7 to 10 years after participation in the initial study of fluconazole prophylaxis for prevention of fungal colonization and infection in preterm infants <1000 grams

CONTACTS AND LOCATIONS:
Overall Officials: David Kaufman, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Neonatal Intensive Care Unit, Charlottesville, Virginia, United States